CLINICAL TRIAL: NCT02936531
Title: Mapping Functional Networks of Brain Activity (Brain Network Activation) Based on Analysis of Evoked Response Potential (ERP) Signals and Registration of Posture and Gait-related Data in FMR1 Premutation Carriers and Patients With FXTAS.
Brief Title: Brain Network Activation and Gait and Posture in FXTAS
Acronym: FXTAS-BNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: ElMindA Ltd (Industry)
Responsible Party: Principal Investigator, Dr. Sharon Hassin, Director, Movement Disorders Institute, Sheba Medical Center
Other Study IDs: SHEBA-3490-16-SMC
Record Dates: First submitted 2016-10-15; First posted 2016-10-18 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Fragile X Associated Tremor-ataxia Syndrome; FXTAS
Keywords: evoked response potential; ERP; Brain Network Activation; BNA; Biomarker
MeSH Terms: conditions — Fragile X Tremor Ataxia Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FXTAS: Patients positive for FMR1 premutation and meet diagnostic criteria for FXTAS
- FMR1 premutation asymptomatic: Patients positive for FMR1 premutation and do not meet diagnostic criteria for FXTAS

SUMMARY:
In this study the investigators aim to identify and characterize a potential neurophysiological biomarker by mapping functional networks of brain activity (Brain Network Activation, BNA) based on analysis of evoked response potential (ERP) signals in both asymptomatic FMR1 premutation carriers and in patients with various stages of FXTAS. Additionally correlations will be studied between these BNA scores and demographics (gender, age and disease duration) as well as genetic mutation and clinical scores.

DETAILED DESCRIPTION:
Fragile X-associated tremor/ataxia syndrome (FXTAS) is a progressive, late-onset (>50 years) multisystem neurodegenerative disorder, associated with an expansion in the 5ʹuntranslated region of the fragile X mental retardation 1 (FMR1) gene that consists of 55-200 CGG repeats, termed the FMR1 gene premutation. While the prevalence of the premutation is 1 in 150-300 females, and 1 in 400-850 males, the penetrance of FXTAS in male carriers is ~40% compared to less than 20% in females.

The mean age of onset of FXTAS is 60 years, presenting with intention tremor, cerebellar ataxia, neuropathic pain, memory and/or executive function deficits, parkinsonism, and psychiatric manifestations such as depression, anxiety and/or apathy.

There are typical MRI findings in FXTAS patients, including increased T2-weighted signal intensity in the middle cerebellar peduncles, cerebellar and cerebral atrophy and volume loss of the corpus callosum.

Currently, no definitive diagnostic tests exist for the symptomatic condition, FXTAS, in FMR1 premutation carriers, making it difficult to diagnose, particularly in the early stages of disease pathology. ElMindA, an Israeli company established in 2006, that focuses on the mapping of neuro-electrophysiological activity, has developed a novel method of mapping functional networks of brain activity (Brain Network Activation or BNA) based on analysis of evoked response potential (ERP) signals. Patients whose underlying disease involves impairment in brain circuitry and connectivity are expected to produce abnormal activity templates in response to the same paradigm, both as a result of failing to adhere to the normal pattern and of recruiting compensatory pathways and strategies to tackle the task. The essence of BNA analysis is the extraction of brain activity patterns common to a group of normal subjects, against which the brain activity of individual subjects may be compared. Patients with FXTAS have been found to exhibit executive and memory deficits along with altered prefrontal cortex activity in functional MRI studies and the investigators suspect that patients with FXTAS and also FMR1 premutation carriers in the early phase of neurodegeneration (even before exhibiting overt clinical symptoms of FXTAS) may display abnormal BNA patterns. Accordingly, at Sheba medical center the investigators have computed individual BNA scores for 30 healthy control subjects and thus defined the BNA patterns of healthy subjects to be used for comparison wit study subjects.

The goal of the study is to identify and characterize a potential neurophysiological biomarker for early stage FXTAS and for disease progression by evaluating the electrophysiological activity in both asymptomatic FMR1 Premutation carriers and in patients with various stages (duration) of FXTAS. Additionally correlations will be studied between these BNA data and demographics (gender, age and disease duration). length of the pathological CGG repeat expansion as well as FXTAS score, gait and posture abnormalities (obtained by instrumental timed up and go evaluation) and neuropsychological status.

Characterization of neuro-electrophysiological biomarkers may be important to detect early transformation from asymptomatic carriership to neurodegeneration and FXTAS and to enable early interventions and monitoring of response to treatment

ELIGIBILITY:
Inclusion Criteria:

* FMR1 premutation carriers (55-200 CGG repeats)
* symptomatic (with possible or probable FXTAS) or neurologically asymptomatic.

Exclusion Criteria:

* Severe disability unable to perform tests
* treatment with neuroleptics
* other brain disease or pathology
* deafness or blindness

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women above the age of 50, that are FMR1 premutation carriers (55-200 CGG repeats), both symptomatic (with possible or probable FXTAS) or neurologically asymptomatic.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
BNA SCORE | 1 day

SECONDARY OUTCOMES:
FXTAS SCORE | 1 day
  Clinical rating scale
Posture and gait data | 1 day
  Posture and gait data from Instrumental" timed up and go" test and items from the FXTAS rating scale.
NeuroTrax™ Computerized Cognitive Tests | 1 day
  Neuropsychological test
MoCA score | 1 day
  Neuropsychological test

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Hassin, MD, Principal Investigator — Movement Disorders Instuitute, Sheba Medical Center
Locations (1):
- Movement Disorders Institute, Sheba Medical center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Leehey MA, Berry-Kravis E, Goetz CG, Zhang L, Hall DA, Li L, Rice CD, Lara R, Cogswell J, Reynolds A, Gane L, Jacquemont S, Tassone F, Grigsby J, Hagerman RJ, Hagerman PJ. FMR1 CGG repeat length predicts motor dysfunction in premutation carriers. Neurology. 2008 Apr 15;70(16 Pt 2):1397-402. doi: 10.1212/01.wnl.0000281692.98200.f5. Epub 2007 Dec 5. PMID 18057320
- [Background] Hagerman RJ, Leehey M, Heinrichs W, Tassone F, Wilson R, Hills J, Grigsby J, Gage B, Hagerman PJ. Intention tremor, parkinsonism, and generalized brain atrophy in male carriers of fragile X. Neurology. 2001 Jul 10;57(1):127-30. doi: 10.1212/wnl.57.1.127. PMID 11445641
- [Background] Hagerman PJ, Hagerman RJ. The fragile-X premutation: a maturing perspective. Am J Hum Genet. 2004 May;74(5):805-16. doi: 10.1086/386296. Epub 2004 Mar 29. PMID 15052536
- [Background] Jacquemont S, Hagerman RJ, Leehey M, Grigsby J, Zhang L, Brunberg JA, Greco C, Des Portes V, Jardini T, Levine R, Berry-Kravis E, Brown WT, Schaeffer S, Kissel J, Tassone F, Hagerman PJ. Fragile X premutation tremor/ataxia syndrome: molecular, clinical, and neuroimaging correlates. Am J Hum Genet. 2003 Apr;72(4):869-78. doi: 10.1086/374321. Epub 2003 Mar 12. PMID 12638084
- [Background] Jacquemont S, Farzin F, Hall D, Leehey M, Tassone F, Gane L, Zhang L, Grigsby J, Jardini T, Lewin F, Berry-Kravis E, Hagerman PJ, Hagerman RJ. Aging in individuals with the FMR1 mutation. Am J Ment Retard. 2004 Mar;109(2):154-64. doi: 10.1352/0895-8017(2004)1092.0.CO;2. PMID 15000674
- [Background] Rogers C, Partington MW, Turner GM. Tremor, ataxia and dementia in older men may indicate a carrier of the fragile X syndrome. Clin Genet. 2003 Jul;64(1):54-6. doi: 10.1034/j.1399-0004.2003.00089.x. PMID 12791039
- [Background] Hall DA, Howard K, Hagerman R, Leehey MA. Parkinsonism in FMR1 premutation carriers may be indistinguishable from Parkinson disease. Parkinsonism Relat Disord. 2009 Feb;15(2):156-9. doi: 10.1016/j.parkreldis.2008.04.037. Epub 2008 Jun 20. PMID 18565783
- [Background] Brunberg JA, Jacquemont S, Hagerman RJ, Berry-Kravis EM, Grigsby J, Leehey MA, Tassone F, Brown WT, Greco CM, Hagerman PJ. Fragile X premutation carriers: characteristic MR imaging findings of adult male patients with progressive cerebellar and cognitive dysfunction. AJNR Am J Neuroradiol. 2002 Nov-Dec;23(10):1757-66. PMID 12427636
- [Background] Grigsby J, Brega AG, Leehey MA, Goodrich GK, Jacquemont S, Loesch DZ, Cogswell JB, Epstein J, Wilson R, Jardini T, Gould E, Bennett RE, Hessl D, Cohen S, Cook K, Tassone F, Hagerman PJ, Hagerman RJ. Impairment of executive cognitive functioning in males with fragile X-associated tremor/ataxia syndrome. Mov Disord. 2007 Apr 15;22(5):645-50. doi: 10.1002/mds.21359. PMID 17266074
- [Background] Ray S, Miller M, Karalunas S, Robertson C, Grayson DS, Cary RP, Hawkey E, Painter JG, Kriz D, Fombonne E, Nigg JT, Fair DA. Structural and functional connectivity of the human brain in autism spectrum disorders and attention-deficit/hyperactivity disorder: A rich club-organization study. Hum Brain Mapp. 2014 Dec;35(12):6032-48. doi: 10.1002/hbm.22603. Epub 2014 Aug 13. PMID 25116862
- [Background] Karalunas SL, Fair D, Musser ED, Aykes K, Iyer SP, Nigg JT. Subtyping attention-deficit/hyperactivity disorder using temperament dimensions: toward biologically based nosologic criteria. JAMA Psychiatry. 2014 Sep;71(9):1015-24. doi: 10.1001/jamapsychiatry.2014.763. PMID 25006969
- [Background] O'Keefe JA, Robertson-Dick E, Dunn EJ, Li Y, Deng Y, Fiutko AN, Berry-Kravis E, Hall DA. Characterization and Early Detection of Balance Deficits in Fragile X Premutation Carriers With and Without Fragile X-Associated Tremor/Ataxia Syndrome (FXTAS). Cerebellum. 2015 Dec;14(6):650-62. doi: 10.1007/s12311-015-0659-7. PMID 25763861
- [Background] Michel CM, Thut G, Morand S, Khateb A, Pegna AJ, Grave de Peralta R, Gonzalez S, Seeck M, Landis T. Electric source imaging of human brain functions. Brain Res Brain Res Rev. 2001 Oct;36(2-3):108-18. doi: 10.1016/s0165-0173(01)00086-8. PMID 11690607
- [Background] Caviness JN, Adler CH, Hentz JG, Shill HA, Evidente VG, Driver-Dunckley ED, Sabbagh MN, Sue L, Beach TG. Incidental Lewy body disease: electrophysiological findings suggesting pre-clinical Lewy body disorders. Clin Neurophysiol. 2011 Dec;122(12):2426-32. doi: 10.1016/j.clinph.2011.03.033. Epub 2011 May 26. PMID 21616709